CLINICAL TRIAL: NCT07281183
Title: The Effects Of Reformer Pilates And Manual Therapy On Pain, Kinesiophobia, Range Of Motion, Quality Of Life, Muscle Strength, Muscle Flexibility And Muscle Shortness In Women With Chronic Low Back Pain
Brief Title: Reformer Pilates and Manual Therapy in Women With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Muhammed Fatih Kavak, Assistant Professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61351342/020-977
Record Dates: First submitted 2025-09-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Pilates Exercise
Keywords: pain; low back; pilates; exercise
MeSH Terms: conditions — Low Back Pain; Pain; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Techniques Group ( MTG ) (Active Comparator): Within the scope of MTG's treatment program; during the first 20 minutes of the session, Transcutaneous Electrical Nerve Stimulation (TENS) was applied to the lumbar region with three channels and a total of six electrodes, while infrared therapy was simultaneously combined and applied to the same region. Soft tissue and mobilization techniques were applied to the lumbar region and surrounding tissues for 15 minutes. Cupping massage and cupping therapy were performed for 5 minutes. Soft tissue mobilization with the Graston technique was applied for 5 minutes, and during the last 5 minutes of the session, a portable percussion massage device was used.
  Interventions: Other: Manual and Physiotherapy Techniques
- MTRPG ( Manual Techniques and Reformer Pilates Group ) (Experimental): In the treatment program of the MTRPG group, in addition to the treatment protocol applied in the MTG group, a reformer Pilates exercise program was implemented. Within this program, the session began with the Footwork series as a 5-10 minute warm-up. Subsequently, the exercises included the running exercise, frog exercise, leg circle series (up-down, circle, one leg side stretch), arm circle exercise series, pelvic lift, elephant exercise, and side stretch mermaid exercise, each performed for 10-15 repetitions. The final 5 minutes of the 50-minute reformer Pilates session consisted of child's pose and spinal stretching series.
  Interventions: Other: Manual and Physiotherapy Techniques and Reformer Pilates Group

INTERVENTIONS:
Other: Manual and Physiotherapy Techniques — Within the scope of MTG's treatment program, during the first 20 minutes of the session, Transcutaneous Electrical Nerve Stimulation (TENS) was applied to the lumbar region with three channels and a total of six electrodes, simultaneously combined with infrared therapy applied to the same area. Soft tissue and mobilization techniques were applied to the lumbar region and surrounding tissues for 15 minutes. Cupping massage and cupping therapy were performed for 5 minutes. The Graston technique was applied for 5 minutes to achieve soft tissue mobilization, and the final 5 minutes of the session were carried out using a portable percussion massage device.
  Arms: Manual Techniques Group ( MTG )
Other: Manual and Physiotherapy Techniques and Reformer Pilates Group — n the treatment program of the MTRPG group, in addition to the treatment protocol applied in the MTG group, a reformer Pilates exercise program was implemented. Within this program, the session began with the Footwork series as a 5-10 minute warm-up. Subsequently, the exercises included the running exercise, frog exercise, leg circle series (up-down, circle, one leg side stretch), arm circle exercise series, pelvic lift, elephant exercise, and side stretch mermaid exercise, each performed for 10-15 repetitions. The final 5 minutes of the 50-minute reformer Pilates session consisted of child's pose and spinal stretching series.
  Arms: MTRPG ( Manual Techniques and Reformer Pilates Group )

SUMMARY:
The purpose of this study is to compare the effects of manual therapy alone and manual therapy combined with Reformer Pilates exercises in women with chronic low back pain (CLBP).

DETAILED DESCRIPTION:
The aim of this study was to compare the effects of manual techniques alone and manual techniques combined with Reformer Pilates exercises in women with chronic low back pain (CLBP), focusing on pain, kinesiophobia, range of motion (ROM), muscle strength, trunk endurance, functional level, and quality of life.

A total of 40 women with CLBP who applied to the Kayroterapi Exercise Center were included. Participants were randomized by odd and even numbers into two groups. The control group (MTG) received a manual techniques protocol once a week for 50 minutes over 8 weeks, while the experimental group (MTRPG) received the same protocol in addition to two 50-minute Reformer Pilates sessions per week. Sociodemographic data were collected through a questionnaire specifically designed for the study. Pain was assessed using the Visual Analog Scale (VAS), kinesiophobia with the Tampa Scale of Kinesiophobia (TSK), and functional disability with the Functional Low Back Pain Scale and the Oswestry Disability Index. Muscle strength was evaluated using manual muscle testing, ROM with a goniometer, and trunk endurance with the sit-and-reach test.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 55 years
* Female gender
* Voluntary participation in the study
* History of low back pain lasting longer than 12 weeks and diagnosis of mechanical low back pain (chronic low back pain)
* No contraindications to exercise
* No physical or mental condition preventing participation in the study

Exclusion Criteria:

* Age below 5 years or above 55 years
* Low back pain lasting less than 12 weeks
* Presence of chronic comorbid disease (e.g., hypertension, diabetes, or other systemic conditions)
* Regular use of medication
* Presence of a neurological pathology
* Any contraindication to exercise
* Inability to establish verbal or visual communication
* Pregnancy

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 40 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-07-19 (Actual); Study Completion 2025-07-19 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity (Visual Analog Scale) | 4 months
  The Visual Analog Scale (VAS), used to assess pain intensity, is a simple, reliable, and easily applicable method. This scale consists of a standard 10 cm vertical or horizontal straight line, with one end indicating "no pain" (0) and the other end indicating "the most severe pain" (10). The patient is asked to mark a point on the line that best represents their current level of pain. The score is then determined based on the location of the mark. Studies have reported that the VAS is a reliable tool for measuring pain intensity.
Oswestry Disability Index: ODI | 4 months
  This scale, which is widely used to assess the level of functional disability in individuals with low back pain, evaluates daily living activities. It consists of a total of 10 subcategories: pain intensity, degree of pain variation, personal care, lifting, sitting, standing, sleeping, social life, traveling, and sexual activity. Each section contains six statements scored from 0 to 5. The individual is asked to choose the statement that best describes their current condition. The total score ranges from 0 to 50. The interpretation of scores is as follows:
  1-10 points: Mild functional disability 11-30 points: Moderate functional disability 31-50 points: Severe functional disability The Turkish validity and reliability study of the scale was conducted by Yakut et al.
Back Pain Functional Scale : FBAS | 4 months
  This scale is used to assess the extent to which individuals' functional levels are affected by low back pain. The functional areas included in the scale are as follows: work, school, home activities, hobbies, forward bending, putting on shoes or socks, lifting objects from the floor, sleeping, sitting, standing, walking, climbing stairs, and driving. For individuals who do not drive, the last item is answered as "traveling."
  Each item is scored between 0 and 5. According to the scoring system:
  (0): Unable to perform the activity
  1. : Extremely difficult
  2. : Very difficult
  3. : Moderately difficult
  4. : Slightly difficult
  5. : Not difficult The total score ranges from 0 to 60. A score of 60 indicates that the individual can perform all activities without any difficulty.
Sit and Reach Test : SRT | 4 months
  It is a simple and widely used physical assessment test designed to evaluate an individual's level of flexibility. During the test, the individual sits on the floor with both legs extended straight and the soles of the feet placed against a box. A 26 cm ruler is placed on top of the box prepared for the measurement. The participant is asked to reach forward as far as possible without bending the knees. The farthest point reached is held for approximately 2 seconds, and the distance is recorded. The best result from two trials is taken and recorded in centimeters.
Range of Motion : ROM | 4 months
  Goniometric measurement is an objective method used in clinical settings to assess normal joint range of motion. During the measurement, the patient is positioned comfortably and appropriately for the joint being evaluated. Before beginning the assessment, the procedure is explained to the patient. All joints are aligned according to the anatomical position, and measurements are taken based on the zero starting position.
  Joint movements are generally assessed within a range of motion from 0° to 180°. Normal range of motion values for the upper and lower extremities and the vertebral column may vary depending on the reference source. In clinical practice, the most commonly used reference standards are those published by Kendall and the American Academy of Orthopaedic Surgeons (AAOS).
Manual Muscle Testing : MMT | 4 months
  It is a clinical method used to assess muscle strength. The basis of these tests was developed by Dr. Robert W. Lovett, Professor of Orthopedics at Harvard Medical School, and was first applied in 1912. The evaluation is scored between 0 and 5 based on the muscle's performance against gravity. The interpretation of these scores may vary depending on the specific muscle being tested.
  5 (Normal): The muscle completes full range of motion against gravity and maximal external resistance.
  4 (Good): The muscle completes full range of motion against gravity but with less than maximal resistance.
  3 (Fair): The muscle completes full range of motion against gravity but without any added resistance.
  2 (Poor): The muscle completes full range of motion in a gravity-eliminated position.
  1 (Trace): Muscle contraction is palpable, but no joint movement occurs. 0 (Zero): No muscle contraction is felt or observed.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Fatih Kavak, Assistant Professor, Study Director — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Design
Supporting Information: Study Protocol